CLINICAL TRIAL: NCT03203538
Title: Effects of Bright Light Intervention for Adaptation to Night Work: Shift Work Simulation Experiments
Brief Title: Light Intervention for Adaptation to Night Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Glamox (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 270755
Record Dates: First submitted 2017-05-03; First posted 2017-06-29 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2018-02

CONDITIONS: Shift-Work Related Sleep Disturbance; Sleep Deprivation; Sleep
Keywords: night work; shift work; light; bright light; sleep; cognitive performance; circadian rhythm
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Three related night shift studies have been planned. Each study investigates how different lighting conditions, administered through LED-based bright light integrated standard room lighting, affects adaptation to simulated night shifts and re adaptation to a day oriented schedule.
  In each study, 28 participants (84 in total) will be exposed to the interventions (light conditions) in a randomized, blinded, controlled, crossover study.
  The simulated night shifts will last from 11pm to 7am. The specific light conditions will last from 11pm to 5am (study 1: 1000 lux vs. 100 lux; study 2: 7000 K vs. 2500 K; study 3: 455 nm vs. 615 nm) where after (from 5am to 7am) all participants will be exposed to the same light conditions (200 lux, 4000 K). After completion of one bout of night work (three consecutive shifts for study 1 and 2; one night shift for study 3) there will be a washout period of four weeks before the participants cross over.
Who Masked: Participant
Masking Description: Participants will not be given information on the hypotheses/ expected effects from the different interventions (light conditions).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Light intensity, 1000 lux (4000 K) (Experimental): Participants will work three consecutive simulated night shifts under full-spectrum LED-light, 1000 lux (4000 Kelvin) administered through standard room lighting.
  Interventions: Device: LED-light, 1000 lux
- Light intensity, 100 lux (4000 K) (Active Comparator): Participants will work three consecutive simulated night shifts under full-spectrum LED-light, 100 lux (4000 Kelvin) administered through standard room lighting.
  Interventions: Device: LED-light, 100 lux
- Colour temperature, 7000 Kelvin (Experimental): Participants will work three consecutive simulated night shifts under full-spectrum LED-light, 7000 K (200 lux) administered through standard room lighting.
  Interventions: Device: LED-light, 7000 K
- Colour temperature, 2500 Kelvin (Active Comparator): Participants will work three consecutive simulated night shifts under full-spectrum LED-light, 2500 K (200 lux) administered through standard room lighting.
  Interventions: Device: LED-light, 2500 K
- Blue light, 455 nm (Experimental): Participants work one night shift with blue LED-light (peak wavelength 455 nm) administered through standard room lighting.
  Interventions: Device: Blue LED-light
- Red light, 615 nm (Active Comparator): Participants work one night shift with red LED-light (peak wavelength 615 nm) administered through standard room lighting.
  Interventions: Device: Red LED-light

INTERVENTIONS:
Device: LED-light, 1000 lux — Full-spectrum light, 1000 lux, 4000 K. Represent a light intensity within acceptable range (light that is not too glary); 4000 K is among the most commonly used indoor light colour temperatures.
  Arms: Light intensity, 1000 lux (4000 K)
Device: LED-light, 100 lux — Full-spectrum light, 100 lux, 4000 K. Represent a light intensity within acceptable range (light that provides sufficient eye sight); 4000 K is among the most commonly used indoor light colour temperatures.
  Arms: Light intensity, 100 lux (4000 K)
Device: LED-light, 7000 K — Full-spectrum light, 7000 K, 200 lux. Represent the upper border of common colour indoor light temperature, 200 lux is a common indoor light intensity.
  Arms: Colour temperature, 7000 Kelvin
Device: LED-light, 2500 K — Full-spectrum light, 2500 K, 200 lux. Represent the lower border of common colour indoor light temperature, 200 lux is a common indoor light intensity.
  Arms: Colour temperature, 2500 Kelvin
Device: Blue LED-light — Blue light with peak wavelength 455 nm. Known to delay the circadian rhythm, suppress melatonin, and increase alertness.
  Arms: Blue light, 455 nm
Device: Red LED-light — Red light with peak wavelength 615 nm. Known not to affect the circadian rhythm, melatonin, and alertness.
  Arms: Red light, 615 nm

SUMMARY:
The project will contribute with new knowledge concerning how aspects of the physical work environment (lighting conditions) can be arranged to facilitate the workers' adaptation to night work. This is important given the reported adverse consequences of shift work for performance, safety, and health. The project involves a series of three experimental, laboratory based shift work simulation studies. The aim is to investigate how different lighting conditions (intensities and colour temperature), administered through light emitting diode (LED) based bright light integrated standard room lighting, affects adaptation to three consecutive simulated night shifts and re adaptation to a day oriented schedule on measures of alertness, cognitive performance, sleep and circadian rhythm. The proposed project examines the effects of interventions that can be applied in naturalistic settings and will be based on new laboratory infrastructure available at the laboratories situated in the Faculty of Psychology, University of Bergen.

DETAILED DESCRIPTION:
Bright light has been suggested as a countermeasure to the negative impact of night work in terms of safety, performance and subsequent sleep. The effect depends on the timing of light (e.g, phase-response curve), duration of light exposure and the intensity of light, as well as the wavelengths that are emitted. Exposure to bright light (more intense than typical room lightning), at evening and night, has been effective in delaying the circadian rhythm to sufficiently adapt to night work both in simulated night work, and in field studies of workers. Blue light has significantly stronger phase shifting effects than other wavelengths of the visible spectrum. The effect of light on the circadian system is mediated by retinal photoresponsive cell population (intrinsically photoresponsive retinal ganglion cells; ipRGC) that contains the photopigment melanopsin, highly sensitive to blue light. These cells signal directly to the suprachiasmatic nuclei (SCN) of the hypothalamus, the circadian pacemaker. Bright light has also been reported to improve alertness and performance during night shifts.

To the best of the investigators knowledge, no shift work simulation study has made the full advance of LED-technology in terms of using light administered via standard room lighting on adaptation to night work. Today, new LED-technology represents an excellent opportunity to study this as roof mounted LED-sources integrated as standard indoor lightening can be programmed to provide a wide range of light intensities and colour temperatures. LED-sources have the advantage over standard light therapy that subjects can be exposed to the therapy via standard room lightening (not confined to a special therapy lamp) thereby allowing the workers to conduct work tasks as normal during light exposure.

Against this backdrop this project aims to investigate how different lighting conditions, administered through LED-based bright light integrated standard room lighting, affects adaptation to three consecutive simulated night shifts and re adaptation to a day oriented schedule on measures of alertness, cognitive performance, sleep and circadian rhythm. In addition, measures of mood, appetite, heart rate variability (HRV), pain sensitivity, moral reasoning, and inflammatory markers will be examined. The researchers also aim to investigate the effects of two extreme monochromatic light conditions (blue vs. red) based on integrated standard room lighting on the adaptation to one simulated night shift.

Study participants will work simulated night shifts (11:00 pm to 07:00 am) in a light laboratory where light parameters (intensity and colour temperature) can be manipulated via roof mounted LED-sources integrated as standard indoor lightening. Participants will be recruited among students at the University of Bergen, and a screening will be done to ensure healthy participants fit for the study. The included participants will take part in experiments with two bouts of three consecutive simulated night shifts (6 nights in total).

HRV will be measured throughout the night shift, and five times, approx. every 1.5 hour (11:30 pm, 01:00 am, 02:30 am, 04:00 am, 05:30 am), the subjects will be tested on a test battery of cognitive tests and will rate their subjective sleepiness. Sleep will be assessed by sleep diary and actigraphy 3 days prior to, during, and 3 days following the shifts. One day before the night shift and the day after the night shift period the circadian rhythm will be measured by saliva samples for estimation of dim light melatonin onset. Prior to-, during- and after the night shifts, participants will undergo a pain sensitivity test. Blood spot samples will be collected at the beginning and the end of each night shift for analysis of inflammatory markers (e.g. interleukins).

ELIGIBILITY:
Inclusion Criteria:

* Participants are physical and mentally healthy (assessed with BMI and 'General Health Questionnaire-12')
* Participants accept to comply with the protocol (refrain from alcohol, tobacco and coffee, and retain regular bed- and wake-times the week before the simulated night shifts)

Exclusion Criteria:

* Neurological, psychiatric or sleep related disorders ('Bergen Insomnia Scale', 'global sleep assessement questionnaire')
* Extreme 'morningness-eveningness' type ('Horne Östberg morningness eveningness questionnaire')
* Use of medication
* Worked night shifts the last 3 months
* Travelled through more than two time zones the last 3 months

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | 3 nights
  Cognitive performance will be measured using the Psychomotor Vigilance Test (PVT). The PVT measures sustained attention, and is considered the 'gold standard' for assessing the effects of sleep deprivation on cognition. The task will be performed approx. every 1.5h throughout the nightshifts.
Circadian phase | 5 days-nights
  Circadian phase will be measured through assessement of 'Dim Light Melatonin Onset' (DLMO). Saliva samples will be collected every hour in the evening (from 7 pm) to one hour past regular bedtime, one day before the first night shift and the day after the night shift period. Saliva will be analyzed for melatonin, giving an estimate on DLMO.
Sleep | 9 days-nights
  Sleep will be measured objectively using actigraphy

SECONDARY OUTCOMES:
Subjective sleepiness | 3 nights
  Karolinska Sleepiness Scale (KSS) will be used to assess subjective sleepiness throughout the night shifts. KSS is a likert scale ranging from 1-9, where subjects rate their sleepiness. '1' indicates 'extremely alert', '9' indicates 'very sleepy/fighting sleep'.
Self-reported sleep | 9 days-nights
  A sleep diary will be used.
Heart rate variability | 3 nights
  'Heart Rate Variability' will be assessed by using Polar heart rate monitor V800 that will continuously monitor 'HRV' through the night.
Interleukin | 3 nights
  Blood spot samples will be analyzed for interleukins (IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-13)
Granulocyte macrophage colony-stimulating factor (GM-CSF) | 3 nights
  Blood-spot samples will be analyzed for GM-CSF.
Interferon gamma (IFN-gamma) | 3 nights
  Blood-spot samples will be analyzed for IFN-gamma.
Tumor necrosis factor alpha (TNF-a) | 3 nights
  Blood-spot samples will be analyzed for TNF-a
Positive and negative affect | 3 nights
  'Positive and Negative Affect Schedule', will be administered to assess mood.
Pain sensitivity | 3 nights
  By using a handheld pressure algometer, Wagner FPIX Force One, the pressure pain threshold will be measured. The test site will be the trapezius muscle, and the pressure will be increased in steps of 5 N/sec until the participant indicates pain.
Headache and eyestrain | 3 nights
  A 'Headache and Eyestrain Scale' will be used to get subjective measures on how participants perceive the lighting conditions.
Appetite/ food cravings | 3 nights
  Appetite/ food cravings for different food types will be assessed using a visual analogue scale to record response to questions like: "How much would you like to eat xxx right now?"
  A 'Dot-probe test' provides measure of attentional bias towards various food types (pictures)
Working memory | 3 nights
  A 'Working Memory Scanning Task' measure ability to encode and maintain information in working memory
Decision/ response execution | 3 nights
  A 'Two-Choice Numerosity Discrimination Task' measure decision criterion and response execution
Decision/ response inhibition | 3 nights
  A 'Reversal Learning Decision Task' measure ability to adjust choices/ response inhibition
Cognitive control | 3 nights
  A 'Task Switching-Performance Test' measure cognitive control
Planning | 3 nights
  The 'Tower of Hanoi Test' measure planning and sequencing abilities
Moral reasoning | 3 nights
  the 'Defining Issues Test' measure moral reasoning.
Cognitive throughput | 3 nights
  A 'Digit Symbol Substitution Test' will be used as a measure of cognitive throughput
Fine motor skills | 3 nights
  The 'grooved pegboard test' assess fine motor skills through the night shifts
Recognition of emotions | 3 nights
  An 'emotional hexagon test', were participants rate standardized pictures of faces expressing different emotions, measure the ability to discriminate between emotional expressions.
Pupil size | 3 nights
  Pupil size will be measured, using a tobii eyetracker, three times during night shifts. This can provide an objective measure of sleepiness.
Core body temperature | 1-2 nights
  To get a secondary measure of circadian phase, core body temperature will be measured using ingestible temperature capsules.
Leadership evaluation | 2 nights, 1 day
  The 'Multifactor Leadership Questionnaire' will be used to assess participants leadership preferences. The questionnaire will be administered during daytime and during night shifts.
Experiences of perceptual anomalies | 3 nights
  The Cardiff Anomalous Perceptions Scale (CAPS) questionnaire will be administered after the night shifts to assess experiences of hallucinations and perceptual anomalies during night shifts. The questionnaire consists of 32 items/questions regarding perceptual anomalies, e.g. "Do you ever notice that sounds are much louder than they normally would be?", that are answered with 'yes' or 'no'. Adding up the number of 'yes' answers gives the CAPS Total Score ranging from 0 (low) to 32 (high). For each item endorsed, participants rate the item for distress, intrusiveness and frequency, giving three subscales. The rating for subscales goes from 1 (low) to 5 (high). Nonendorsed items are considered to have a score of 0 on subscales. For each subscale the possible range goes from 0 (low) to 160 (high).
Objective sleepiness, sleep and sleep stages | 3 nights and sleep periods
  A subgroup of participants (12-16 in each experiment) will be subject to electroencephalography (EEG) during night shifts, and polysomnography (PSG) after night shifts. EEG will provide a measure of electrical activity in the brain during wakefulness, and can provide an objective measure of sleepiness. PSG will be conducted in the sleep period after night shifts, and allow for the scoring of sleep stages. PSG is considered the gold standard for measuring sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Erlend Sunde, Principal Investigator — University of Bergen, department of psychosocial science
Locations (1):
- The faculty of psychology, University of Bergen, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No
After the project has ended the data will be anonymized and no direct recognizable information will be stored.

REFERENCES:
- [Derived] Sunde E, Harris A, Olsen OK, Pallesen S. Moral decision-making at night and the impact of night work with blue-enriched white light or warm white light: a counterbalanced crossover study. Ann Med. 2024 Dec;56(1):2331054. doi: 10.1080/07853890.2024.2331054. Epub 2024 Apr 18. PMID 38635448
- [Derived] Sunde E, Mrdalj J, Pedersen TT, Bjorvatn B, Gronli J, Harris A, Waage S, Pallesen S. Bright light exposure during simulated night work improves cognitive flexibility. Chronobiol Int. 2022 Jul;39(7):948-963. doi: 10.1080/07420528.2022.2050922. Epub 2022 Mar 28. PMID 35343353
- [Derived] Sunde E, Pedersen T, Mrdalj J, Thun E, Gronli J, Harris A, Bjorvatn B, Waage S, Skene DJ, Pallesen S. Alerting and Circadian Effects of Short-Wavelength vs. Long-Wavelength Narrow-Bandwidth Light during a Simulated Night Shift. Clocks Sleep. 2020 Nov 25;2(4):502-522. doi: 10.3390/clockssleep2040037. PMID 33255613
- [Derived] Sunde E, Pedersen T, Mrdalj J, Thun E, Gronli J, Harris A, Bjorvatn B, Waage S, Skene DJ, Pallesen S. Blue-Enriched White Light Improves Performance but Not Subjective Alertness and Circadian Adaptation During Three Consecutive Simulated Night Shifts. Front Psychol. 2020 Aug 18;11:2172. doi: 10.3389/fpsyg.2020.02172. eCollection 2020. PMID 33013558
- [Derived] Sunde E, Mrdalj J, Pedersen T, Thun E, Bjorvatn B, Gronli J, Harris A, Waage S, Pallesen S. Role of nocturnal light intensity on adaptation to three consecutive night shifts: a counterbalanced crossover study. Occup Environ Med. 2020 Apr;77(4):249-255. doi: 10.1136/oemed-2019-106049. Epub 2020 Feb 4. PMID 32019847